CLINICAL TRIAL: NCT04976348
Title: The Multicenter Cardiology Monitoring Platform Registry (mCMP-registry)
Brief Title: The Multicenter Cardiology Monitoring Platform Registry
Acronym: mCMPregistry
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Zuyderland Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: NL76585.068.21
Record Dates: First submitted 2021-06-22; First posted 2021-07-26 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Cardiomyopathies; Atrial Fibrillation; Ventricular Arrythmia; Coronary Artery Disease; Ventricular Tachycardia
Keywords: heart failure; registry; cardiomyopathy; atrial fibrillation; ventricular tachycardia; coronary artery disease
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Atrial Fibrillation; Coronary Artery Disease; Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — blood, urine, and cardiac biopsy samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Consenting participants: All subjects aged ≥16 years referred to the cardiology or genetic department for heart failure like symptoms (as stated in the ESC 2016 Guidelines) or for cardiac/cardiogenetic screening.

SUMMARY:
The multicenter Cardiology Monitoring Platform registry (mCMP-registry) is a prospective observational registry including multi-omics (diagnostic) measurements performed as part of routine clinical care, bio-banking (optional), and yearly questionnaires (optional).

It's objective is to optimize (early) diagnosis and risk-stratification of (early) cardiovascular diseases, specifically cardiomyopathy phenotypes, arrhythmias, and coronary artery disease, and to create a better understanding of underlying pathophysiological processes.

DETAILED DESCRIPTION:
Rationale: Heart failure (HF) represents a heterogeneous range of clinical overlapping cardiomyopathy phenotypes, resulting from multifactorial environmental insults in the presence or absence of a genetic predisposition. A better understanding of (early) cardiomyopathy phenotypes, related cardiovascular diseases, their underlying pathophysiological processes, and their related disease burden is key to pave the way for novel preventive and/or intervention studies.

Objective: To optimize (early) diagnosis and risk-stratification of (early) cardiovascular diseases, specifically cardiomyopathy phenotypes, arrhythmias, and coronary artery disease, and to create a better understanding of underlying pathophysiological processes.

Study design: The multicenter Cardiology Monitoring Platform registry (mCMP-registry) is an investigator-initiated multicentre prospective observational registry including multi-omics (diagnostic) measurements performed as part of routine clinical care, bio-banking (optional), and yearly questionnaires (optional).

Study population: All subjects aged ≥16 years that have been referred to the cardiology or genetics department for cardiac symptoms, cardiac screening or cardiogenetic screening are eligible for inclusion.

Main study parameters/endpoints: This is a prospective registry from which multiple research questions can be answered. In general, two main approaches will be used: (A) a data-driven (multi-)omics approach which aims to identify clusters of patients to predict clinical outcome, to improve (early) diagnosis, and/or to identify clusters of patients that share underlying pathophysiological processes; (B) a hypothesis-driven approach in which clinical parameters are tested for their (incremental) diagnostic and/or prognostic value.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the cardiology or genetic department for heart failure like symptoms (as stated in the ESC 2016 Guidelines(3)) or for cardiac/cardiogenetic screening;
* Age ≥16 years.

Exclusion Criteria:

* Unwillingness to participate or unable to give written informed consent (e.g. due to language barriers or severe intellectual disability).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects aged ≥16 years that have been referred to the cardiology or genetics department for cardiac symptoms, cardiac screening or cardiogenetic screening are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2051-12 (Estimated); Study Completion 2051-12 (Estimated)

PRIMARY OUTCOMES:
(sudden) cardiac death or heart transplantation | through study completion, an average of 15 years
  Death attributed to a cardiac cause or sudden, or heart transplantation.

SECONDARY OUTCOMES:
Heart Failure hospitalization | through study completion, an average of 15 years
  Hospitalization due to cardiac decompensation or prolonged hospitalization due to cardiac decompensation
Life-threatening arrhythmias | through study completion, an average of 15 years
  justified implantable cardioverter-defibrillator shock, justified anti-tachypacing therapy, cardiac arrest, hemodynamic unstable ventricular tachycardia
Quality of life EQ-5D questionnaire | through study completion, an average of 15 years
  EQ-5D questionnaire
Economic burden | through study completion, an average of 15 years
  institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire (iPCQ) and iMTA Medical Consumption Questionnaire (iMCQ)

OTHER OUTCOMES:
Age | through study completion, an average of 15 years
  Age based on birth date
Sex | through study completion, an average of 15 years
  Sex (biological)
Body mass index | through study completion, an average of 15 years
  BMI
Underlying pathogenic | through study completion, an average of 15 years
  variants found in cardiac associated genes
Medication usage | through study completion, an average of 15 years
  Prescribed medication

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Peter Brunner-La Rocca, Prof., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Henkens MTHM, Weerts J, Verdonschot JAJ, Raafs AG, Stroeks S, Sikking MA, Amin H, Mourmans SGJ, Geraeds CBG, Sanders-van Wijk S, Barandiaran Aizpurua A, Uszko-Lencer NHMK, Krapels IPC, Wolffs PFG, Brunner HG, van Leeuwen REW, Verhesen W, Schalla SM, van Stipdonk AWM, Knackstedt C, Li X, Abdul Hamid MA, van Paassen P, Hazebroek MR, Vernooy K, Brunner-La Rocca HP, van Empel VPM, Heymans SRB. Improving diagnosis and risk stratification across the ejection fraction spectrum: the Maastricht Cardiomyopathy registry. ESC Heart Fail. 2022 Apr;9(2):1463-1470. doi: 10.1002/ehf2.13833. Epub 2022 Feb 4. PMID 35118823
- See also: Website with more information on the study — http://cardiomyopathyresearch.eu